CLINICAL TRIAL: NCT06320483
Title: Evaluation of the Effectiveness and Safety of Vibro-acoustic Pulmonary Therapy (VAPT) in Complex Therapy for Acute Respiratory Failure of Mixed Type I-II Stages in Comparison With Percussion Massage in Cardiac Surgical Patients in the Early Postoperative Period
Status: Recruiting | Type: Observational
Sponsor: Bark Technology LLP (Industry)
Responsible Party: Sponsor
Other Study IDs: BT-01-23
Record Dates: First submitted 2023-10-04; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Surgical Patients (CABG,Mammary Coronary Bypass Surgery,Plastic and Replacement of Valves, Atrial Septal Defect,Ventricular Septal Defect)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group with percussion massage
- Group with vibroacoustic massage
  Interventions: Device: Vibroacoustic device BARK VibroLUNG

INTERVENTIONS:
Device: Vibroacoustic device BARK VibroLUNG — The BARK VibroLUNG vibroacoustic device is intended for the treatment and prevention of respiratory pathologies.
  The BARK VibroLUNG vibroacoustic device with accessories is a medical device and is intended for the treatment of pathological conditions associated with obstructive and restrictive lung diseases in patients in medical institutions.
  Field of application: physiotherapy of the chest organs, treatment and prevention of respiratory failure.
  The therapeutic mechanism of action is due to three main effects: improved bronchial drainage, improved ventilation-perfusion ratios, and the "lung opening" maneuver.
  Groups: Group with vibroacoustic massage

SUMMARY:
The goal of this observational study is to evaluate the effectiveness and safety of vibro-acoustic pulmonary therapy (VAPT) in complex therapy for the acute respiratory failure of mixed type I-II stages in comparison with percussion massage in cardiac surgical patients in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years to 80 years inclusive
* Body mass index from 18.5 to 35
* Physical status according to ASA II to ASA III (inclusive)
* Performed planned cardiac surgery (CS) under general anaesthesia with tracheal intubation and mechanical ventilation lasting more than 3 hours using a heart-lung machine (no more than 120 minutes)
* Left ventricular injection fraction before surgical treatment is above 40%
* Development of postoperative mixed ARF grade 1-2 (clinical criteria). SpO2 less than 95% with FiO2 21%.
* Stable-severe condition of the patient according to vital signs:

  1. stable hemodynamics (norepinephrine and/or adrenaline less than 0.15 mcg/kg/min, and/or dobutamine less than 10 mcg/kg/min, and/or no need for vasopressin (ADH) for 6 hours or more)
  2. absence of acute kidney injury (urine output more than 500 ml/day)
  3. stable respiratory dynamics.P/F more than 150 units, SpO2 more than 70% with FiO2 21%.Tracheal extubation within 8 hours of completion of surgery
  4. absence of critical coagulopathy (platelets more than 50 units/l)
  5. absence of acute cerebral insufficiency (GCS more than 12 points)
  6. absence of acute liver failure (bilirubin less than 30 units/l)
* Relieved postoperative pain syndrome and delirium (NRS less than 5 points, BPS less than 6 points, CAM-ICU (-), RASS -3-0 points).

Exclusion Criteria:

* The presence of implanted or external medical electronic-mechanical devices in the impact projection (pacemaker, circulatory support devices, etc.);
* Severe hypocoagulation, risk of hematoma formation or bleeding in the projection of exposure;
* Severe hypercoagulation, risk of formation and/or migration of blood clots or emboli along the great vessels in the projection of exposure;
* Acute cerebrovascular accident (ACB), first 1-3 days;
* Cerebral Edema;
* High intracranial pressure;
* The presence of many purulent or burn wound surfaces in the projection of exposure;
* Presence of an unstable rib fracture;
* Pneumohemomediastinum and/or subcutaneous emphysema of the chest;
* Risk of development of hemo-pneumothorax;
* Osteomyelitis of the ribs and/or thoracic spine;
* Spinal fracture without orthopedic fixation;
* Trauma to the chest or abdomen with bleeding;
* High risk of seizures (CNS pathologies);
* The presence of an oncological process in the projection of exposure with destruction of tumor tissue and the risk of bleeding and/or metastasis;
* The presence of endothoracic and/or large endovascular implants (aortic stents, intra-aortic balloon pumps, endocardial catheters, mechanical heart valves, vena cava filters, subcutaneous venous ports, permanent hemodialysis devices);
* Heart rhythm disturbances (ventricular fibrillation, ventricular tachycardia);
* Hypovolemia;
* Disturbances of water-electrolyte balance and acid-base balance;
* Meningoencephalitis;
* Destructive purulent pneumonia;
* High risk of pulmonary hemorrhage;
* Hiatal hernia;
* Risk of dislocation of implanted drainage tubes and catheters;
* The presence of multiple wound surfaces in the projection of exposure;
* Severe bullous deformation of the lungs;
* Severe kyphoscoliosis;
* Spontaneous pneumothorax within the last year;
* Estimated systolic pressure over the pulmonary artery more than 50 mm Hg. Art.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes from 18 to 80 years old who are undergoing planned hospitalization for cardiac surgery (CABG, Mammary Coronary Bypass Surgery, Plastic and Replacement of Valves, Atrial Septal Defect, Ventricular Septal Defect)
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Partial pressure of oxygen (PaO2) | on days 2 and 3
Partial pressure of carbon dioxide (PaCO2) | on days 2 and 3
Blood oxygen saturation level (SpO2) on pulse oximeter (peripheral capillary oxygenation) | on days 2,3,4,5,6,7
Ratio of peripheral arterial oxygen saturation(SaO2) to the inspired fraction of oxygen FiO2 | on days 2 and 3
Ratio of venous saturation (SvO2) to the inspired fraction of oxygen FiO2 | on days 2,3,4,5,6,7
ROX Index | on days 2 and 3
P/F index (ratio of arterial blood PO2 to oxygen fraction) | on days 2 and 3

SECONDARY OUTCOMES:
pH of blood | on days 2 and 3
BE (base excess) of blood | on days 2 and 3
CBC indicators (hemoglobin) | on days 2,3,4,5,6,7 for hemoglobin
CBC indicators (hematocrit) | on days 2 and 3 for hematocrit
CBC indicators (platelets) | on days 2 and 3 for platelets
Coagulogram indicators (prothrombin time) | on days 2 and 3
Coagulogram indicators (prothrombin index) | on days 2 and 3
Coagulogram indicators (international normalized ratio) | on days 2 and 3
Coagulogram indicators (fibrinogen) | on days 2 and 3
Coagulogram indicators (activated partial thromboplastin time) | on days 2 and 3
Number of days spent in the high dependency unit (intensive care ward in the department) | through study completion, an average of 7days
Number of days in hospital | through study completion,an average of 7days
Number of days of O2 support | through study completion,an average of 7days
Proportion of patients with postoperative complications (pneumonia/atelectasis/pulmonary infiltration) | through study completion,an average of 7days

CONTACTS AND LOCATIONS:
Locations (5):
- Kazakhstan (5):
  - JSC "National Research Cardiac Surgery Center", Astana
  - State-owned public enterprise with the right of economic management "Atyrau Regional Cardiology Center", Atyrau
  - State-owned public enterprise with the right of economic management "Regional Cardiology Center", Oral
  - State-owned public enterprise with the right of economic management "Pavlodar Regional Cardiology Center", Pavlodar
  - State-owned public enterprise with the right of economic management "East Kazakhstan Regional Hospital", Ust-Kamenogorsk